CLINICAL TRIAL: NCT06693141
Title: Comparison of the Effects of Erector Spinae Plane Block and Intrathecal Morphine Administration on Intraoperative Sevoflurane Consumption in Disc Surgeries
Brief Title: Effects of Erector Spinae Plane Block and Intrathecal Morphine Administration on Intraoperative Sevoflurane Consumption
Status: Not yet recruiting | Type: Observational
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Yusuf Özgüner, Principal Investigator, Ankara Etlik City Hospital
Other Study IDs: Bengü Tez
Record Dates: First submitted 2024-11-15; First posted 2024-11-18 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Postoperative Pain; Anesthesia
Keywords: Erector Spinae Plane block; Intrathecal morphine
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ESP: ESP block was applied to patients in this group in the preoperative period.
  Interventions: Other: ESP block
- ITM: Intrathecal morphine was applied to patients in this group in the preoperative period.
  Interventions: Other: ITM
- Control: Patients who did not undergo ESP block or ITM were included in this group.

INTERVENTIONS:
Other: ESP block — ESP block was applied to the patients.
  Groups: ESP
Other: ITM — ITM was applied to the patients.
  Groups: ITM

SUMMARY:
In our study, the investigators aimed to compare the intraoperative sevoflurane consumption and postoperative analgesic needs of patients who underwent lumbar disc herniation surgery and received either ESP block or ITM in the preoperative period with a control group.

DETAILED DESCRIPTION:
The amount of volatile anesthetic agents used for anesthesia maintenance can be significantly reduced with potent and long-acting analgesic interventions administered during the preoperative period. Such interventions enable the maintenance of anesthesia with more optimal levels of agents during surgery, providing significant advantages in terms of both patient safety and cost.

Studies have recommended multimodal analgesia approaches involving the Erector Spinae Plane (ESP) block and intrathecal morphine (ITM) injection for various surgical procedures. These two methods, through different mechanisms of action, not only reduce intraoperative anesthetic agent consumption but also play a critical role in postoperative pain management. Although studies have investigated the effects of ESP block and ITM injection on intraoperative volatile anesthetic consumption, there is limited research directly comparing their impacts on volatile anesthetic consumption and postoperative analgesic requirements.

In our study, we aimed to compare the intraoperative sevoflurane consumption and postoperative analgesic needs of patients who underwent lumbar disc herniation surgery and received either ESP block or ITM in the preoperative period with a control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years
* Patients receiving general anesthesia
* Patients with an ASA score of I-II
* Patients undergoing elective surgery for single-level lumbar disc herniation
* Patients who provided informed consent after being informed

Exclusion Criteria:

Patients who did not provide informed consent after being informed

* Patients over 65 years of age
* Patients with an ASA score of III or higher
* Patients with recurrent lumbar disc herniation (LDH)
* Patients undergoing surgery for multi-level LDH
* Patients with a body mass index (BMI) of 30 or higher
* Patients with allergies to morphine or bupivacaine
* Patients with major cardiac, respiratory, hepatic, renal, neurological, or psychiatric diseases
* Patients with a history of alcohol or substance abuse
* Patients with a local infection at the injection site
* Patients with bleeding diathesis
* Patients with a history of anticoagulant medication use
* Patients with contraindications to spinal or regional anesthesia

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients operated for single level and non-recurring lumbar disc herniation.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Estimated)
Dates: Start 2024-11-20 (Estimated); Primary Completion 2025-01-10 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
Intraoperative Sevoflurane consumption | 60 minutes after anesthesia induction
  End-expiratory sevoflurane concentration was monitored every 5 minutes for 60 minutes. The mean sevoflurane concentration in the first 60 minutes was calculated.

SECONDARY OUTCOMES:
Rescue analgesic consumption | 2 hours postoperatively
  When numerical rating scale was 4 or above, rescue analgesic was administered to the patient.
Rescue analgesic consumption | 4 hours postoperatively
  When numerical rating scale was 4 or above, rescue analgesic was administered to the patient.
Rescue analgesic consumption | 8 hours postoperatively
  When numerical rating scale was 4 or above, rescue analgesic was administered to the patient.
Rescue analgesic consumption | 12 hours postoperatively
  When numerical rating scale was 4 or above, rescue analgesic was administered to the patient.
Rescue analgesic consumption | 24 hours postoperatively
  When numerical rating scale was 4 or above, rescue analgesic was administered to the patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Ankara, Varlık Mahallesi, Halil Sezai Erkut Caddesi Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yorukoglu HU, Icli D, Aksu C, Cesur S, Kus A, Gurkan Y. Erector spinae block for postoperative pain management in lumbar disc hernia repair. J Anesth. 2021 Jun;35(3):420-425. doi: 10.1007/s00540-021-02920-0. Epub 2021 Mar 22. PMID 33751203
- [Background] Lal A, Singh MK, Kanaujia SK, Mishra NK, Singh BP, Singh GP. Comparison of Intrathecal Morphine Versus Erector Spinae Plane Block for Perioperative Analgesia in Patients Undergoing Lumbar Spine Surgery: A Randomized Control Trial. Cureus. 2024 Jul 17;16(7):e64775. doi: 10.7759/cureus.64775. eCollection 2024 Jul. PMID 39156461
- [Result] Nashibi M, Sezari P, Safari F, Teymourian H, Asgari S, Mottaghi K. The effect of erector spinae plane block on the use of anesthetic medications in lumbar spine surgery. Agri. 2023 Oct;35(4):228-235. doi: 10.14744/agri.2022.48992. PMID 37886866